CLINICAL TRIAL: NCT00942591
Title: Efficacy, Safety and Tolerability of Atorvastatin 40 mg in Patients With Relapsing-remitting Multiple Sclerosis Treated With Interferon-beta-1b.SWiss Atorvastatin and Interferon-Beta 1b Trial In Multiple Sclerosis.
Brief Title: Atorvastatin 40 mg in Patients With Relapsing-Remitting Multiple Sclerosis Treated With Interferon-Beta-1b
Acronym: SWABIMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: PharmaPart (Industry); Laboratory: Viollier AG Spalenring 145 / 147 Postfach 4002 Basel (Unknown)
Responsible Party: Prof. Heinrich Paul Mattle, Chefarzt, Department of Neurology, University Hospital Bern, Freiburgstr. 3010 Bern
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17/05; CWCNS01
Record Dates: First submitted 2009-07-17; First posted 2009-07-21 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; interferon beta; atorvastatin
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b; Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Interferon beta-1b AND atorvastatin
  Interventions: Drug: Interferon beta 1b; Drug: Atorvastatin
- 2 (Active Comparator): Interferon beta-1b
  Interventions: Drug: Interferon beta 1b

INTERVENTIONS:
Drug: Interferon beta 1b
Drug: Atorvastatin
  Arms: 1

SUMMARY:
Title: Efficacy, safety and tolerability of Atorvastatin 40 mg in patients with relapsing-remitting multiple sclerosis treated with interferon-beta-1b SWiss Atorvastatin and Interferon-Beta 1b Trial In Multiple Sclerosis

Short title: "SWABIMS"

Study phase: Phase IIb study

Study design: Multi-center, randomized, rater-blinded, parallel-group-study in Switzerland

Investigational product: Atorvastatin 40mg every day (oral) plus Interferon-beta

Reference product: Interferon-beta-1b 250mg given

Indication: Relapsing-remitting multiple sclerosis (RR-MS)

Study objectives: Comparison of efficacy, safety and tolerability of combination of Atorvastatin 40mg (per os) daily and Interferon-beta-1b e.o.d in patients with relapsing-remitting multiple sclerosis compared to monotherapy with Interferon-beta-1b e.o.d.

Primary Endpoint: Proportion of patients with new T2 lesions after 15 months of treatment.

DETAILED DESCRIPTION:
Background

Multiple sclerosis is considered to be a chronic inflammatory demyelinating autoimmune disease of the central nervous system. Statins are lipid-lowering drugs which inhibit the 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA-) reductase, which is the main regulatory enzyme of cholesterol biosynthesis. In recent years many studies have demonstrated, that statins have anti-inflammatory and immunomodulatory properties in addition to their lipid-lowering effects. Therefore, statins seem to have therapeutic potential in immune-mediated disorders such as multiple sclerosis. Studies in experimental allergic encephalomyelitis (EAE), the animal model for the human demyelinating disease multiple sclerosis, as well as smaller studies in patients with relapsing-remitting multiple sclerosis showed beneficial effect on the course of the disease. But there are also reports of negative impact of statins on multiple sclerosis. Therefore, bigger studies are needed to investigate the therapeutical potential of statins in multiple sclerosis.

Objective

The objectives of this study are to assess the efficacy, safety and tolerability of the combination of Atorvastatin 40mg p.o. daily and Interferon-beta-1b sc e.o.d compared to monotherapy with Interferon-beta-1b sc e.o.d in patients with relapsing-remitting multiple sclerosis.

Methods

Multi-center, rater-blinded, parallel-group, two arm, randomized study. Patients with relapsing-remitting forms of MS, respecting all inclusion/exclusion criteria, will be randomized into two equal-size parallel arms after three months of treatment with Interferon-beta-1b, receiving Atorvastatin 40mg/d or not. Enrolment of 80 patients (1/2 in the Atorvastatin group) is planned. Patients providing written informed consent will be treated for 15 months.

Inclusion criteria: Patients with relapsing-remitting forms of multiple sclerosis with disease duration > 3 month and < 5 years, at least 1 relapse in the past two years, > 3 Lesions on spinal or brain-MRI, EDSS score between 0 and 3.5, inclusive, age between 18 and 55 years.

Exclusion criteria: Any disease other than multiple sclerosis that would better explain the patient's signs and symptoms, Primary progressive MS, Secondary progressive MS, and others.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing-remitting forms of multiple sclerosis (according to McDonald's criteria)
* At least 1 relapse in the past two year
* > 3 Lesions on spinal or brain-MRI
* EDSS score between 0 and 3.5, inclusive
* Age between 18 and 55 years
* Written informed consent
* Negative pregnancy test results (all women)

Exclusion Criteria

* Any disease other than multiple sclerosis that would better explain the patient's signs and symptoms
* Primary progressive MS
* Secondary progressive MS
* Uncontrolled severe medical disorder
* A history of drug abuse in the 6 months prior to screening
* Previous therapy with Monoclonal antibodies, mitoxantrone, cytotoxic or immunosuppressive therapy (except steroids)
* Participation in any other studies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2005-05; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with new T2 lesions on MRI. | 15 months

SECONDARY OUTCOMES:
Gd-enhancing lesion on T1-weighted images | 15 months
Clinical disease progression | 15 months
Time to first relapse | 15 months
Cortical atrophy | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Mattle, Principal Investigator — Dep. of Neurology, Bern University hospital
Locations (1):
- Prof. H. Mattle, Dep. of Neurology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Paty DW, Li DK; UBC MS/MRI Study Group and IFNB Multiple Sclerosis Study Group. Interferon beta-lb is effective in relapsing-remitting multiple sclerosis. II. MRI analysis results of a multicenter, randomized, double-blind, placebo-controlled trial. 1993 [classical article]. Neurology. 2001 Dec;57(12 Suppl 5):S10-5. No abstract available. PMID 11902589
- [Background] Youssef S, Stuve O, Patarroyo JC, Ruiz PJ, Radosevich JL, Hur EM, Bravo M, Mitchell DJ, Sobel RA, Steinman L, Zamvil SS. The HMG-CoA reductase inhibitor, atorvastatin, promotes a Th2 bias and reverses paralysis in central nervous system autoimmune disease. Nature. 2002 Nov 7;420(6911):78-84. doi: 10.1038/nature01158. PMID 12422218
- [Background] Kwak B, Mulhaupt F, Myit S, Mach F. Statins as a newly recognized type of immunomodulator. Nat Med. 2000 Dec;6(12):1399-402. doi: 10.1038/82219. PMID 11100127
- [Derived] Kamm CP, Mattle HP; SWABIMS Study Group. SWiss Atorvastatin and interferon Beta-1b trial In Multiple Sclerosis (SWABIMS)--rationale, design and methodology. Trials. 2009 Dec 14;10:115. doi: 10.1186/1745-6215-10-115. PMID 20003436